CLINICAL TRIAL: NCT06185569
Title: FREnch Data on Outcomes in HR+/HER2- Early Breast Cancer Patients With oncotypeDX Recurrence Score-guided Therapy
Brief Title: FREDO-ODX Study: FREnch Data on Outcomes in HR+/HER2- Early Breast Cancer Patients With oncotypeDX Recurrence Score-guided Therapy
Acronym: FREDO-ODX-23
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/804
Record Dates: First submitted 2023-10-16; First posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Early breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to assess the clinical outcomes in real-life setting of early breast cancer RH+ HER2- patients with systemic therapy guided by Oncotype DX (ODX) Breast Recurrence Score®.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old With invasive breast carcinoma diagnosed on biopsy or surgical sample (histological evidence) Operable breast cancer HR+ (at least ER+) /HER2- tumors With ODX assay performed

Exclusion Criteria:

* Inoperable tumor(s) or inoperable patient (e.g., patient too frail to undergo surgery) Synchronous breast cancers with different clinico-pathological features (e.g. : HR+/HER2 negative and triple-negative or HER2-positive breast cancer Patient undergoing neoadjuvant chemotherapy or neoadjuvant hormone therapy Nodal involvement in more than 4 lymph nodes (pN2 or higher) Metastatic breast cancer at diagnosis Other malignancy diagnosed in the past 10 years (except for cutaneous malignancies other than melanoma) The patient participated in the RxPONDER study in France The patient communicated a refusal to participate in the study (via a refusal letter to the investigator) Legal incapacity or limited legal capacity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥ 18 years old, with invasive breast carcinoma diagnosed on biopsy or surgical sample (histological evidence), Operable breast cancer HR+ (at least ER+) /HER2- tumors with ODX assay performed
Sampling Method: Non-Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2023-10-15 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
to evaluate the clinical outcomes represented by iDFS in French early breast cancer patients with Oncotype DX (ODX) Breast Recurrence Score® (RS) results-guided therapy | time between surgery and recurrence (local, regional, distant), contralateral breast cancer, second cancer or death (all causes), whichever occurs first, assessed up to 5 years

SECONDARY OUTCOMES:
Breast cancer-specific survival | time between surgery and death related to breast cancer, assessed up to 5 years
Distant disease-free survival | time between surgery and distant recurrence or death (all causes), whichever occurs first, assessed up to 5 years
Locoregional relapse-free survival | time between surgery and progression/recurrence (local, regional), ipsilateral DCIS or death (all causes), whichever occurs first, assessed up to 5 years
Overall Survival | time between surgery and death, assessed up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Elsa CURTIT, Principal Investigator — Centre Hospitalier Universitaire de Besancon
Locations (5):
- France (5):
  - CHU Besançon, Besançon
  - Clinique Tivoli Ducos, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - AP-HP - Hôpital Tenon, Paris
  - Centre Catalan d'Oncologie, Perpignan

IPD SHARING:
Plan to Share IPD: No